CLINICAL TRIAL: NCT02421861
Title: Critical Care Anxiety and Long-Term Outcomes Management
Acronym: CALM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Jennifer Jutte, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 48493-G
Record Dates: First submitted 2015-04-10; First posted 2015-04-21 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Anxiety
Keywords: anxiety; intensive care unit; critical care
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Anxiety Management (AM) (Experimental)
  Interventions: Behavioral: Anxiety Management in the ICU
- Usual Care (UC) (Placebo Comparator)
  Interventions: Other: Usual Care (UC)

INTERVENTIONS:
Behavioral: Anxiety Management in the ICU — The AM intervention is based on a Cognitive-Behavioral Therapy (CBT) approach, empirically supported in other settings, though we do not know whether this approach will be effective for ICU patients. It will offer all participants core aspects of CBT including: (1) establish rapport/therapeutic alliance; (2) anxiety psychoeducation; (3) normalization of difficulties; (4) establishment of a sense of hope; (5) reflective listening; (6) supportive statements; (7) exposure to anxious thoughts/feelings; (8) directive statements; and (9) provision of coping strategies. It will consist of modules that include the aforementioned core aspects and "optional" modules based on each participant's anxiety experience and preference.
  Arms: Anxiety Management (AM)
Other: Usual Care (UC) — The UC group will receive usual care as per the Harborview Medical Center usual care standard. Because this is an effectiveness trial, treatment decisions for UC participants will be left to the discretion of the primary provider and/or primary medical team and may or may not include: (1) referral to rehab psychology C&L service; (2) referral to psychiatry C&L service; or (3) pharmacologic management.
  Arms: Usual Care (UC)

SUMMARY:
The aims of this study are to (1) test the benefits of a non-pharmacologic anxiety management approach with patients who are critically ill and/or traumatically injured during intensive care hospitalization and (2) test whether this approach reduces anxiety and improves engagement in rehabilitation therapies, shortens duration of hospitalization, and improves psychological and quality of life outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Ability to read, write, and speak English
* Alert (Best RASS ICU sedation score ≥-2)
* Current CAM-ICU test negative
* Expected ICU stay ≥48 hours
* Anxiety Visual Analog Scale (VAS-A) score ≥30
* Prescribed rehabilitation therapy at eligibility

Exclusion Criteria:

* Inability to communicate (verbally, or via hand writing/gestures)
* Greater than 90% probability of mortality in hospital
* Anticipated discharge to hospice or transition to end-of-life care
* Pre-existing cognitive impairment (e.g., dementia, pervasive developmental disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Anxiety (Visual Analog Scale for Anxiety (VAS-A) | Participants will be followed for the duration of hospitalization, an expected average of 13 days and not more than 45 days
  Anxiety at discharge and change in anxiety from baseline to discharge as measured by the Visual Analog Scale for Anxiety (VAS-A)

SECONDARY OUTCOMES:
Engagement in rehabilitation therapies (As measured by a 2-item engagement questionnaire) | As measured by a 2-item engagement questionnaire (developed specifically for this study) at the time of hospital discharge (i.e., based on an expected average duration of hospitalization of 13 days and not more than 45 days)
Length of ICU and Hospital Stay | Measured in days (an expected average ICU stay=5 days and average Hospital stay=13 days and not more than 45 days)
Long-Term Anxiety and Depressive Symptoms (as measured by the Hospital Anxiety and Depression Scale (HADS) | 3 months after enrollment as measured by the Hospital Anxiety and Depression Scale (HADS)
Long-Term Posttraumatic Stress Symptoms (as measured by the PCL-5) | 3 months after enrollment as measured by the PCL-5
Health-Related Quality of Life (as measured by the EQ-5D-5L and SF-36) | 3 months after enrollment